CLINICAL TRIAL: NCT00458029
Title: Studies to Treat Or Prevent Pediatric Type 2 Diabetes (STOPP-T2D) Middle-School Based Primary Prevention Trial (HEALTHY)
Brief Title: Middle-School Based Primary Prevention Trial of Type 2 Diabetes
Acronym: HEALTHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U01DK061230-HEALTHY; U01DK061230 (NIH); U01DK061223 (NIH); U01DK061231 (NIH); U01DK061249 (NIH)
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes risk factors; obesity; prevention; adolescence; school based
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- School based intervention (Experimental): Integration of activities, events, and programs affecting total school food service environment, physical education class, behavior change, promotion, and communications
  Interventions: Behavioral: integrated program of nutrition, activity, behavior, and promotion
- Control (No Intervention): Observational control

INTERVENTIONS:
Behavioral: integrated program of nutrition, activity, behavior, and promotion — implemented across 5 half-year periods: winter/spring 2007, fall 2007, winter/spring 2007, fall 2008, winter/spring 2008
  Arms: School based intervention

SUMMARY:
HEALTHY was a primary prevention trial conducted in 42 middle schools at 7 locations across the US to impact risk factors for type 2 diabetes in adolescents. Students were recruited at start of 6th grade (fall 2006) and followed to end of 8th grade (spring 2009). Half of the schools were randomized to receive an intervention that integrated four components: the school nutrition environment, physical education class activities, behavior change initiatives, and educational and promotional communications activities.

DETAILED DESCRIPTION:
In response to increases in incident cases of type 2 diabetes in American children and youth, NIDDK funded a multi-site primary prevention trial designed to moderate risk for type 2 diabetes in middle school aged children. In pilot studies, it was found that an indicator of adiposity, a body mass index greater than the 85th percentile for gender and age, was the most prevalent, modifiable risk factor for diabetes in this age group. In addition, indicators of insulin resistance and dysglycemia, elevated mean fasting insulin and glucose levels, were assessed to determine if the intervention was capable of reducing these risk factors for diabetes in middle school aged children.

The trial was conducted at 7 field centers in 42 middle schools randomly assigned to intervention or control. Following student recruitment and baseline data collection in the first semester of 6th grade (2006), the intervention was implemented in the second semester of 6th grade (2007) and continued throughout 7th (school year 2007-2008) and 8th (school year 2008-2009) grades. All students were exposed to components of the intervention, which were implemented school-wide or grade-wide; however, only students who provided appropriate informed consent and assent participated in data collection and evaluation. The primary objective of the trial was to determine if, at the end of the 8th grade, the intervention significantly impacted the risk for developing type 2 diabetes compared to control.

Six pilot studies were performed to collect data to guide the development of an intervention. The prior studies focused on:

* Establishing the feasibility of recruiting students and obtaining physical and physiological measurements, including fasting and 2-hour post glucose load blood draws (early 2003).
* Evaluating a physical education (PE) class program designed to increase moderate-to-vigorous physical activity (late 2003).
* Testing the ability of a nutrition intervention to change food and beverage offerings in school food service and vending (early 2004).
* Implementing a program that integrated the PE class and food service nutrition interventions with a communications and awareness campaign (fall 2004).
* Determining the feasibility of a behavior change intervention, delivered through in-class and other school settings and family outreach, to accomplish self monitoring and goal setting (fall 2005).
* Evaluating PE class activities targeting 7th and 8th graders and a training and support program to motivate PE teacher buy-in and adherence (fall 2005).

Formative research was conducted to inform the creation of all intervention components.

Based on a comprehensive review of the literature and the pilot study results, a robust multi-component intervention was developed to impact the environment and lifestyle choices of middle school children. The intervention consisted of the following integrated components:

* changes in the nutritional quality of food and beverage offerings throughout the total school food environment, including cafeteria meals and programs, a la carte, and vending machines;
* changes in the physical education (PE) program, equipment, and teacher training to increase both participation and number of minutes spent in moderate-to-vigorous physical activity when implemented by PE teachers in PE class;
* brief classroom activities designed to increase knowledge, enhance decision making skills, promote peer involvement and interaction, and enhance social influence;
* individual and group behavior change initiatives aimed at promoting healthier behaviors through self monitoring, goal setting, and problem solving;
* family outreach to involve parents/guardians and family members by providing information and strategies to support youth in accomplishing behavioral goals; and
* school-wide communications to enhance and promote changes in nutrition, activity, and behavior.

In addition to the primary objective of affecting risk for T2D, major secondary objectives were to: further understand and characterize the etiology of risk of T2D in this age group; evaluate the ability of the intervention to influence lifestyle changes and choices both in and out of school; determine the cost-effectiveness of the intervention; compare academic performance, attendance, and comportment in intervention versus control schools; and describe the influence of non-study changes in the school environment that affect student nutrition and physical activity. Finally, data were collected to evaluate the degree to which the components of the intervention were delivered and administered as planned.

ELIGIBILITY:
Inclusion Criteria:

* Middle school student body is at least 50% minority (defined as African American, Hispanic/Latino, and/or Native American) and/or greater than 50% eligible for free or reduced lunch.
* Middle school annual school-wide attrition from all causes is <= 25% (estimate determined from data provided by the school).
* Middle school expected cohort size at end of study is at least 50 per school determined by applying 50% anticipated enrollment rate and annual school-wide attrition rate over 3 years.
* Student able to participate in the school's standard PE program.
* Student's parent/guardian has provided informed consent for the child to participate in data collection and evaluation procedures.
* Student has provided informed assent to participate in data collection and evaluation procedures.

Exclusion Criteria: (none specified)

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4603 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) >= 85th percentile, adjusted for gender and age | baseline, end of 7th grade, end of study
Fasting glucose (mg/dL) | baseline, end of study
Fasting insulin (mU/mL) | baseline, end of study

SECONDARY OUTCOMES:
Lipids (total cholesterol, HDL, LDL, triglycerides) | baseline, end of study
Other laboratory indicators of diabetes and obesity risk, such as HbA1c | baseline, end of study
Blood pressure | baseline, end of study
Waist circumference | baseline, end of study
Physical activity | baseline, end of study
Sedentary behavior | baseline, end of study
Fitness | baseline, end of study
Daily nutritional intake | baseline, end of study
PE class activity level (MVPA by heart rate monitor) | baseline, end of 7th grade, end of study
Quality-adjusted life years saved (QALYS) | baseline, end of 7th grade, end of study
Total school food environment amounts and nutrients | baseline, end of 7th grade, end of study
Grade and school level state standardized test score pass rates | end of 6th, 7th, 8th grades
Grade and school level attendance rates | end of 6th, 7th, 8th grades
Grade and school level comportment rates (i.e., referral to administrative offices for disciplinary action) | end of 6th, 7th, 8th grades
Costs associated with intervention delivery and administration | once per intervention semester (5 x)
Decisions, policies, and activities at the school, local, state, or federal level that influence the school environment for nutrition and physical activity | once per year (3 x)

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Foster, PhD, Principal Investigator — Temple University; Kathryn Hirst, PhD, Principal Investigator — George Washington University Biostatistics Center
Locations (8):
- United States (8):
  - University of California at Irvine, Irvine, California
  - George Washington University Biostatistics Center, Rockville, Maryland
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/healthy/?query=healthy
URL: https://repository.niddk.nih.gov/studies/healthy/?query=healthy

REFERENCES:
- [Background] HEALTHY Study Group; Hirst K, Baranowski T, DeBar L, Foster GD, Kaufman F, Kennel P, Linder B, Schneider M, Venditti EM, Yin Z. HEALTHY study rationale, design and methods: moderating risk of type 2 diabetes in multi-ethnic middle school students. Int J Obes (Lond). 2009 Aug;33 Suppl 4(Suppl 4):S4-20. doi: 10.1038/ijo.2009.112. PMID 19623188
- [Background] Drews KL, Harrell JS, Thompson D, Mazzuto SL, Ford EG, Carter M, Ford DA, Yin Z, Jessup AN, Roullet JB; HEALTHY Study Group. Recruitment and retention strategies and methods in the HEALTHY study. Int J Obes (Lond). 2009 Aug;33 Suppl 4(Suppl 4):S21-8. doi: 10.1038/ijo.2009.113. PMID 19623184
- [Background] Gillis B, Mobley C, Stadler DD, Hartstein J, Virus A, Volpe SL, El ghormli L, Staten MA, Bridgman J, McCormick S; HEALTHY Study Group. Rationale, design and methods of the HEALTHY study nutrition intervention component. Int J Obes (Lond). 2009 Aug;33 Suppl 4(Suppl 4):S29-36. doi: 10.1038/ijo.2009.114. PMID 19623185
- [Background] McMurray RG, Bassin S, Jago R, Bruecker S, Moe EL, Murray T, Mazzuto SL, Volpe SL; HEALTHY Study Group. Rationale, design and methods of the HEALTHY study physical education intervention component. Int J Obes (Lond). 2009 Aug;33 Suppl 4(Suppl 4):S37-43. doi: 10.1038/ijo.2009.115. PMID 19623187
- [Background] Venditti EM, Elliot DL, Faith MS, Firrell LS, Giles CM, Goldberg L, Marcus MD, Schneider M, Solomon S, Thompson D, Yin Z; HEALTHY Study Group. Rationale, design and methods of the HEALTHY study behavior intervention component. Int J Obes (Lond). 2009 Aug;33 Suppl 4(Suppl 4):S44-51. doi: 10.1038/ijo.2009.116. PMID 19623189
- [Background] DeBar LL, Schneider M, Ford EG, Hernandez AE, Showell B, Drews KL, Moe EL, Gillis B, Jessup AN, Stadler DD, White M; HEALTHY Study Group. Social marketing-based communications to integrate and support the HEALTHY study intervention. Int J Obes (Lond). 2009 Aug;33 Suppl 4(Suppl 4):S52-9. doi: 10.1038/ijo.2009.117. PMID 19623190
- [Background] Schneider M, Hall WJ, Hernandez AE, Hindes K, Montez G, Pham T, Rosen L, Sleigh A, Thompson D, Volpe SL, Zeveloff A, Steckler A; HEALTHY Study Group. Rationale, design and methods for process evaluation in the HEALTHY study. Int J Obes (Lond). 2009 Aug;33 Suppl 4(Suppl 4):S60-7. doi: 10.1038/ijo.2009.118. PMID 19623191
- [Result] Baranowski T, Cooper DM, Harrell J, Hirst K, Kaufman FR, Goran M, Resnicow K; STOPP-T2D Prevention Study Group. Presence of diabetes risk factors in a large U.S. eighth-grade cohort. Diabetes Care. 2006 Feb;29(2):212-7. doi: 10.2337/diacare.29.02.06.dc05-1037. PMID 16443862
- [Result] Jago R, Harrell JS, McMurray RG, Edelstein S, El Ghormli L, Bassin S. Prevalence of abnormal lipid and blood pressure values among an ethnically diverse population of eighth-grade adolescents and screening implications. Pediatrics. 2006 Jun;117(6):2065-73. doi: 10.1542/peds.2005-1716. PMID 16740849
- [Result] Cullen KW, Hartstein J, Reynolds KD, Vu M, Resnicow K, Greene N, White MA; Studies to Treat or Prevent Pediatric Type 2 Diabetes Prevention Study Group. Improving the school food environment: results from a pilot study in middle schools. J Am Diet Assoc. 2007 Mar;107(3):484-9. doi: 10.1016/j.jada.2006.12.004. PMID 17324667
- [Result] Hartstein J, Cullen KW, Reynolds KD, Harrell J, Resnicow K, Kennel P; STOPP T2D Prevention Study Group. Impact of portion-size control for school a la carte items: changes in kilocalories and macronutrients purchased by middle school students. J Am Diet Assoc. 2008 Jan;108(1):140-4. doi: 10.1016/j.jada.2007.10.005. PMID 18156001
- [Result] Studies to Treat or Prevent Pediatric Type 2 Diabetes Prevention Study Group. Prevalence of the metabolic syndrome among a racially/ethnically diverse group of U.S. eighth-grade adolescents and associations with fasting insulin and homeostasis model assessment of insulin resistance levels. Diabetes Care. 2008 Oct;31(10):2020-5. doi: 10.2337/dc08-0411. Epub 2008 Jun 30. PMID 18591405
- [Result] Jago R, Baranowski T, Watson K, Bachman C, Baranowski JC, Thompson D, Hernandez AE, Venditti E, Blackshear T, Moe E. Development of new physical activity and sedentary behavior change self-efficacy questionnaires using item response modeling. Int J Behav Nutr Phys Act. 2009 Mar 31;6:20. doi: 10.1186/1479-5868-6-20. PMID 19335875
- [Result] Jago R, McMurray RG, Bassin S, Pyle L, Bruecker S, Jakicic JM, Moe E, Murray T, Volpe SL. Modifying middle school physical education: piloting strategies to increase physical activity. Pediatr Exerc Sci. 2009 May;21(2):171-85. doi: 10.1123/pes.21.2.171. PMID 19556623
- [Result] HEALTHY Study Group; Kaufman FR, Hirst K, Linder B, Baranowski T, Cooper DM, Foster GD, Goldberg L, Harrell JS, Marcus MD, Trevino RP. Risk factors for type 2 diabetes in a sixth- grade multiracial cohort: the HEALTHY study. Diabetes Care. 2009 May;32(5):953-5. doi: 10.2337/dc08-1774. Epub 2009 Feb 5. PMID 19196888
- [Result] Baranowski T, Watson KB, Bachman C, Baranowski JC, Cullen KW, Thompson D, Siega Riz AM. Self efficacy for fruit, vegetable and water intakes: Expanded and abbreviated scales from item response modeling analyses. Int J Behav Nutr Phys Act. 2010 Mar 29;7:25. doi: 10.1186/1479-5868-7-25. PMID 20350316
- [Result] HEALTHY Study Group; Foster GD, Linder B, Baranowski T, Cooper DM, Goldberg L, Harrell JS, Kaufman F, Marcus MD, Trevino RP, Hirst K. A school-based intervention for diabetes risk reduction. N Engl J Med. 2010 Jul 29;363(5):443-53. doi: 10.1056/NEJMoa1001933. Epub 2010 Jun 27. PMID 20581420
- [Result] Jago R, Drews KL, McMurray RG, Thompson D, Volpe SL, Moe EL, Jakicic JM, Pham TH, Bruecker S, Blackshear TB, Yin Z. Fatness, fitness, and cardiometabolic risk factors among sixth-grade youth. Med Sci Sports Exerc. 2010 Aug;42(8):1502-10. doi: 10.1249/MSS.0b013e3181d322c4. PMID 20139783
- [Result] Marcus MD, Baranowski T, DeBar LL, Edelstein S, Kaufman FR, Schneider M, Siega-Riz AM, Staten MA, Virus A, Yin Z. Severe obesity and selected risk factors in a sixth grade multiracial cohort: the HEALTHY study. J Adolesc Health. 2010 Dec;47(6):604-7. doi: 10.1016/j.jadohealth.2010.04.017. Epub 2010 Jun 29. PMID 21094439
- [Result] Siega-Riz AM, El Ghormli L, Mobley C, Gillis B, Stadler D, Hartstein J, Volpe SL, Virus A, Bridgman J; HEALTHY Study Group. The effects of the HEALTHY study intervention on middle school student dietary intakes. Int J Behav Nutr Phys Act. 2011 Feb 4;8:7. doi: 10.1186/1479-5868-8-7. PMID 21294869
- [Derived] Mietus-Snyder M, Drews KL, Otvos JD, Willi SM, Foster GD, Jago R, Buse JB; HEALTHY Study Group. Low-density lipoprotein cholesterol versus particle number in middle school children. J Pediatr. 2013 Aug;163(2):355-62. doi: 10.1016/j.jpeds.2013.01.012. Epub 2013 Feb 14. PMID 23415622
- [Derived] Buse JB, Kaufman FR, Linder B, Hirst K, El Ghormli L, Willi S; HEALTHY Study Group. Diabetes screening with hemoglobin A(1c) versus fasting plasma glucose in a multiethnic middle-school cohort. Diabetes Care. 2013 Feb;36(2):429-35. doi: 10.2337/dc12-0295. Epub 2012 Nov 27. PMID 23193207
- [Derived] Willi SM, Hirst K, Jago R, Buse J, Kaufman F, El Ghormli L, Bassin S, Elliot D, Hale DE; HEALTHY Study Group. Cardiovascular risk factors in multi-ethnic middle school students: the HEALTHY primary prevention trial. Pediatr Obes. 2012 Jun;7(3):230-9. doi: 10.1111/j.2047-6310.2011.00042.x. Epub 2012 Mar 28. PMID 22461375
- [Derived] Marcus MD, Foster GD, El Ghormli L, Baranowski T, Goldberg L, Jago R, Linder B, Steckler A, Trevino R. Shifts in BMI category and associated cardiometabolic risk: prospective results from HEALTHY study. Pediatrics. 2012 Apr;129(4):e983-91. doi: 10.1542/peds.2011-2696. Epub 2012 Mar 19. PMID 22430457
- [Derived] DeBar LL, Schneider M, Drews KL, Ford EG, Stadler DD, Moe EL, White M, Hernandez AE, Solomon S, Jessup A, Venditti EM; HEALTHY study group. Student public commitment in a school-based diabetes prevention project: impact on physical health and health behavior. BMC Public Health. 2011 Sep 20;11:711. doi: 10.1186/1471-2458-11-711. PMID 21933431
- See also: public access to HEALTHY intervention program materials — http://www.healthystudy.org